CLINICAL TRIAL: NCT05387889
Title: Piloting an Evidence-based Mobile Mindfulness Practice to Support Self-management Among Underserved and Racial Minority Adults With Pulmonary Hypertension
Brief Title: Piloting Mindfulness Meditation Program for Underserved Racial Minority Adults With Pulmonary Hypertension
Acronym: MMPH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: State University of New York at Buffalo (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Principal Investigator, Tania T Von Visger, Principal Investigator, State University of New York at Buffalo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12345; UL1TR001412 (NIH)
Record Dates: First submitted 2022-03-25; First posted 2022-05-24 (Actual); Results first posted 2023-11-08 (Actual); Last update posted 2023-11-08 (Actual); Status verified 2023-11

CONDITIONS: Hypertension, Pulmonary
Keywords: pulmonary hypertension; racial minority; complementary health approach; integrative therapy; mindfulness-based intervention; symptom management; health-related quality of life
MeSH Terms: conditions — Hypertension, Pulmonary | interventions — Mindfulness

STUDY DESIGN:
Intervention Model Description: wait-listed control comparative groups
Masking Description: All participants will receive intervention according to the wait-listed control comparative groups. Therefore, masking is not applicable in this study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Arm (Experimental): This treatment Arm will receive MMPH intervention first, while the wait-listed group waits until this group is complete.
  Then the wait-listed group will receive the same intervention after the first group completes it.
  Interventions: Behavioral: Mindfulness Meditation for Pulmonary Hypertension (MMPH)
- Comparison Arm or Waited List Arm (Active Comparator): This active comparator Arm will not receive MMPH intervention at the beginning. They will receive the intervention once the Treatment Group completed the intervention.
  Interventions: Behavioral: Mindfulness Meditation for Pulmonary Hypertension (MMPH)

INTERVENTIONS:
Behavioral: Mindfulness Meditation for Pulmonary Hypertension (MMPH) — Eight weeks of Mindfulness Meditation practice for patients with Pulmonary Hypertension condition. The content will focus on how to apply Mindfulness concepts to the everyday management of symptoms and stress.
  Other Names: MMPH intervention

SUMMARY:
The MMPH program will include two Zoom-delivered sessions (Weeks #1 & #4), six video-recorded sessions (Weeks #2, #3, #5, #6, #7, #8), and daily mindfulness meditation practice using a mobile APP during an eight-week study period. Similar to the Urban Zen Integrative Therapy intervention, each MMPH session will include Gentle Body Movement (GBM,10-min), Restorative Pose (Pose,10-min), and Body Awareness Meditation (BAM, 20-min). Self-guided audio-video modules of various durations will be available according to participants' preference and level of comfort (5, 10, 20 minutes). The mobile-APP content will reinforce Zoom content such as mindful breathing, GBM of upper extremities, GBM of lower extremities, Pose sitting, Pose lying, and BAM practices. The MMPH content will be tailored to health management needs specific to PH with cultural consideration of mindfulness-related concepts (stress, responding to stress, resiliency).

DETAILED DESCRIPTION:
Study design: This study will engage community-dwelling URM adults with PH living in Western New York. We will use a two-group comparative study design where waitlisted participants will serve as controls. Considering a 20% attrition rate in a behavioral health intervention study, we aim to enroll a total of 20, with at least 16 participants to address study aims (8-10 in each group). As a pilot study, power analysis is not necessary. Statistical analysis will include descriptive statistics, mixed-effect modeling for repeated measures, and within-group and between-groups comparisons using t-tests or Wilcoxon signed-rank test as appropriate and Cohen's d effect size calculation. Multi-time data collection will be done via daily mobile-APP use.

Setting/ Sample: We will recruit PH patients from two PH clinics managed by UB PH Specialists, a local PH support group, and through the CTSI community outreach programs. Recruitment materials will be disseminated to PH physicians, PH support group leaders, and community leaders, inviting patients to participate in the study. Interested patients will contact research staff by phone or email and will be guided to complete the eligibility questionnaire online using REDCAP.

If eligible and interested, participants will meet with research staff to provide verbal consent via Zoom after reviewing the Consent Form content. During the meeting, the research staff will review the purpose of the study, study procedures, and risks and benefits. After providing verbal consent, participants will complete the Demographic and Clinical Characteristic questionnaire online. The initial 10 participants enrolled will be scheduled to begin the program, including mutually agreeable Zoom #1 and Zoom #2 appointments. They will also be provided with a de-identified user ID and password to register and download the MMPH APP to his/her personal phone (Table 1- Study Procedure).

Intervention: MMPH program will include two Zoom-delivered sessions (Weeks #1 & #4) and the daily practice of Mindfulness meditation using a mobile-APP for an eight-week study period. Similar to the UZIT intervention, each MMPH session will include Gentle Body Movement (GBM,10-min), Restorative Pose (Pose,10-min), and Body Awareness Meditation (BAM, 20-min). Self-guided audio-video modules of various durations will be available according to participants' preference and level of comfort (5, 10, 20 minutes). The mobile-APP content will reinforce Zoom content such as mindful breathing, GBM of upper extremities, GBM of lower extremities, Pose sitting, Pose lying, and BAM practices. The MMPH content will be tailored to health management needs specific to PH with cultural consideration of mindfulness-related concepts (stress, responding to stress, resiliency).

Individual Zoom Interviews: will take place at a convenient time during the last week of the study. The primary focus of this interview is to collect qualitative data about their participation experience in the MMPH program. Standard qualitative thematic analysis procedures will be employed. The following open-ended questions will guide the discussion: 1) What are your general impressions of the program?; 2) How does this program affect you in the management of your PH-related symptoms?; 3) What do you like & do not like about the program?; and 4) What improvements would you recommend?

ELIGIBILITY:
Inclusion Criteria:

* Adults (>18 years)
* PH confirmed by standard guidelines
* Self-identified as URM person
* Willingness to participate in the mindfulness practice program for the duration of the study period
* Able to ambulate independently
* English-speaking
* Have access to a mobile phone

Exclusion Criteria:

* Known pregnancy
* Have psychiatric conditions requiring hospitalization within the last year
* Current practitioner of mind-body practices
* Current user of Mindfulness APP
* Deaf or hard of hearing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2022-06-17 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2023-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tania Von Visger, Principal Investigator — State University of New York at Buffalo School of Nursing
Locations (1):
- SUNY at Buffalo School of Nursing, Buffalo, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment Arm - Group 1: This treatment Arm will receive MMPH intervention first, while the wait-listed group waits until this group is complete.
  Then the wait-listed group will receive the same intervention after the first group completes it.
  Mindfulness Meditation for Pulmonary Hypertension (MMPH): Eight weeks of Mindfulness Meditation practice for patients with Pulmonary Hypertension condition. The content will focus on how to apply Mindfulness concepts to the everyday management of symptoms and stress.
- Comparison Arm or Waited List Arm - Group 2: This active comparator Arm will not receive MMPH intervention at the beginning. They will receive the intervention once the Treatment Group completed the intervention.
  Mindfulness Meditation for Pulmonary Hypertension (MMPH): Eight weeks of Mindfulness Meditation practice for patients with Pulmonary Hypertension condition. The content will focus on how to apply Mindfulness concepts to the everyday management of symptoms and stress.
Period: Overall Study
Arm/Group | Treatment Arm - Group 1 | Comparison Arm or Waited List Arm - Group 2
Started | 9 | 6
Completed | 9 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment Arm - Group 1 | Comparison Arm or Waited List Arm - Group 2 | Total
Number analyzed (Participants) | 9 | 6 | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 6 | 12
  >=65 years | 3 | 0 | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.00 (13.92) | 47.50 (7.82) | 51.40 (11.97)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 6 | 14
  Male | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 8 | 5 | 13
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 9 | 6 | 15
Depressive symptoms on the 27-point Patient Health Questionnaire-9 Scales [Mean (Standard Deviation); unit: units on a scale] | 6.12500 (5.30330) | 9.80000 (8.55570) | 7.9625 (6.9295)
PH-related Quality of Life on the 50-point EmPHasis-10 Scale [Mean (Standard Deviation); unit: units on a scale] | 22.7500 (11.5357) | 25.6000 (9.7877) | 24.175 (10.6617)
Mindfulness Level on the 40-point Cognitive and Affective Mindfulness Scale [Mean (Standard Deviation); unit: units on a scale] | 28.2500 (4.89168) | 25.8000 (2.28035) | 27.025 (3.586)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Depressive Symptoms on the 27-point Patient Health Questionnaire-9 Scales (PHQ-9) to Week #8.
Description: Patient Health Questionnaire-9 is a validated, self-reported questionnaire assessing depressive symptoms over the past few weeks. Possible scores range from 0 to 27, indicating the levels of depression (0-4 = None or Minimal; 5-9 = Mild; 10-14 = Moderate; 15-19 = Moderately Severe; 20- 27 = Severe).
  Depressive symptoms comparison between Group 1 and Group 2 at the end of the intervention (Week #8).
  Depressive symptoms comparison at Baseline vs. Week #8 within Group 1 participants who received the intervention.
  Depressive symptoms comparison at Baseline vs. Week #8 within Group 2 participants who received the intervention.
Time Frame: Baseline and at the end of the study intervention (Week #8)
Population: For this analysis, 9 patients were analyzed for Arm 1, and 6 patients were analyzed for Arm 2.
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Treatment Arm - Group 1 | Comparison Arm or Waited List Arm - Group 2
Number analyzed (Participants) | 9 | 6
score on scale | 3.44444 (2.403) | 7.6666 (2.011)
Statistical Analysis 1: Comparison: Treatment Arm - Group 1 vs Comparison Arm or Waited List Arm - Group 2; Test type: Superiority; p < 0.054, ANCOVA — The threshold for the level of significance is set at less than or equal to 0.05; Mean Difference (Final Values) = 0.05

2. Secondary Outcome: Change From Baseline in PH-related Quality of Life on the 50-point EmPHasis-10 Scales to Week #8.
Description: EmPHasis-10 (full name, not an abbreviation) is a validated, self-reported standardized questionnaire assessing PH-related quality of life over the past few weeks. The EmPHasis-10 questionnaire is used during clinical assessments to determine how pulmonary hypertension affects someone's life. Possible scores range from 0 to 50, (0 = high quality of life; 50 = poor quality of life)
  Change = (Week #8 Score - Baseline Score)
  Health-related quality of life comparison between Group 1 and Group 2 at the end of the intervention (Week #8).
  Health-related quality of life comparison at Baseline vs. Week #8 within Group 1 participants who received the intervention.
  Health-related quality of life comparison at Baseline vs. Week #8 within Group 2 participants who received the intervention.
Time Frame: Baseline and at the end of the study intervention (Week #8)
Population: For this analysis, 9 patients were analyzed for Arm 1, and 6 patients were analyzed for Arm 2.
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Treatment Arm - Group 1 | Comparison Arm or Waited List Arm - Group 2
Number analyzed (Participants) | 9 | 6
score on scale | 19.0 (11.068) | 23.166 (10.10)
Statistical Analysis 1: Comparison: Treatment Arm - Group 1 vs Comparison Arm or Waited List Arm - Group 2; Test type: Superiority; p < 0.25, ANCOVA — The threshold for the level of significance is set at less than or equal to 0.05; Mean Difference (Final Values) = 0.05

3. Secondary Outcome: Change From Baseline in Mindfulness Level on the 40-point Cognitive and Affective Mindfulness Scale-Revised (CAMS-R) to Week #8.
Description: Cognitive and Affective Mindfulness Scale-Revised (CAMS-R) is a validated, self-reported questionnaire assessing the degree of an individual's Mindfulness Level over the past few weeks. Possible scores range from 10 to 40 (10 = low level of mindfulness; 40 = high level of mindfulness)
  Mindfulness level comparison between Group 1 and Group 2 at the end of the intervention (Week #8).
  Mindfulness level comparison at Baseline vs. Week #8 within Group 1 participants who received the intervention.
  Mindfulness level comparison at Baseline vs. Week #8 within Group 2 participants who received the intervention.
Time Frame: Baseline and at the end of the study intervention (Week #8)
Population: For this analysis, 9 patients were analyzed for Arm 1, and 6 patients were analyzed for Arm 2.
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Treatment Arm - Group 1 | Comparison Arm or Waited List Arm - Group 2
Number analyzed (Participants) | 9 | 6
score on scale | 31.000 (5.567) | 27.00 (4.242)
Statistical Analysis 1: Comparison: Treatment Arm - Group 1 vs Comparison Arm or Waited List Arm - Group 2; Test type: Superiority; p < 0.07, ANCOVA — The threshold for the level of significance is set at less than or equal to 0.05; Mean Difference (Final Values) = 0.05

ADVERSE EVENTS:
Time Frame: 16 weeks
Groups:
- Treatment Arm: This treatment Arm will receive MMPH intervention first, while the wait-listed group waits until this group is complete.
  Then the wait-listed group will receive the same intervention after the first group completes it.
  Mindfulness Meditation for Pulmonary Hypertension (MMPH): Eight weeks of Mindfulness Meditation practice for patients with Pulmonary Hypertension condition. The content will focus on how to apply Mindfulness concepts to the everyday management of symptoms and stress.
Arm/Group | Treatment Arm | Comparison Arm or Waited List Arm
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/6
Other Adverse Events (participants affected / at risk) | 0/9 | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-09-15): https://cdn.clinicaltrials.gov/large-docs/89/NCT05387889/Prot_SAP_000.pdf
  • Informed Consent Form (2022-06-13): https://cdn.clinicaltrials.gov/large-docs/89/NCT05387889/ICF_001.pdf